CLINICAL TRIAL: NCT00208845
Title: Hypernet- Hypertension ED Surveillance
Brief Title: Hypernet- Hypertension Screening
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Debra Houry, MD, MPH, Principal Investigator, Emory University
Other Study IDs: 0996-2001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Asymptomatic Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adult ED patients

SUMMARY:
Identify untreated, asymptomatic hypertension in ER patients

DETAILED DESCRIPTION:
this was a prospective study done with no intervention- the study has since been completed

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic hypertension

Exclusion Criteria:

* cardiac symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ED patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Heilpern, MD, Principal Investigator — Emory University